CLINICAL TRIAL: NCT01252849
Title: A Prospective, Randomized, Controlled Evaluation of Open-Angle Glaucoma Subjects on Two Topical Hypotensive Medications, Implanted With One, Two, or Three Trabecular Micro-Bypass Stents
Brief Title: Purpose of This Study is to Evaluate the Safety and Efficacy of One, Two, or Three iStents for the Reduction of Intraocular Pressure in Open-angle Glaucoma Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCF-016
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: Open angle; Glaucoma; surgery; Glaucoma, Open-Angle; Ocular Hypertension; Eye Diseases
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Intervention Model Description: iStent 1, 2, or 3 stents
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- First Arm: One iStent, medication (Experimental): Device: One iStent, medication
  Interventions: Device: iStent
- Second Arm: Two iStents, medication (Experimental): Device: Two iStent devices, medication
  Interventions: Device: iStent
- Third Arm: Three iStents, medication (Experimental): Device: Three iStent devices, medication
  Interventions: Device: iStent

INTERVENTIONS:
Device: iStent — Implantation of One iStent through a small temporal clear corneal incision.
  Arms: First Arm: One iStent, medication
Device: iStent — Implantation of Two iStents through a small temporal clear corneal incision
  Arms: Second Arm: Two iStents, medication
Device: iStent — Implantation of Three iStents through a small temperal clear corneal incision
  Arms: Third Arm: Three iStents, medication

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the iStent medical device that is implanted into the eye and designed to reduce eye pressure in patients with your condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* Subject on two topical hypotensive medications

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Mean diurnal IOP reduction of greater than or equal to 20% at month 12 vs. baseline | 12 Months

SECONDARY OUTCOMES:
Mean diurnal IOP <18 mmHg at month 12 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- S.V. Malayan's Ophthalmology Centre, Yerevan, Armenia